CLINICAL TRIAL: NCT04381429
Title: Effect of Postprandial Insulin Administration of Faster-acting Insulin Analogue Versus Pre-prandial Administration of Acting-insulin Analogue in Cystic Fibrosis Related Diabetes : MIRE Trial
Brief Title: Effect of Postprandial Insulin Administration of Faster-acting Insulin Analogue Versus Pre-prandial Administration of Acting-insulin Analogue in Cystic Fibrosis Related Diabetes
Acronym: MIRE
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Difficulties of inclusion in this rare pathology
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 7546
Record Dates: First submitted 2020-04-30; First posted 2020-05-08 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Cystic Fibrosis-related Diabetes
MeSH Terms: interventions — Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1: A-F-A-F (Active Comparator): The study is an open, randomized, two-treatment - 4 periods of 3 months - 2 group cross-over superiority study.
  All patients will test both insulin treatments (A and F) in alternating periods.
  The patients of group 1 will start with pre-prandial aspart insulin (NovoRapid).
  Each treatment period will last 3 months.
  Interventions: Drug: A-F-A-F (NovoRapid-FIASP-NovoRapid-FIASP)
- Groupe 2: F-A-F-A (Active Comparator): The study is an open, randomized, two-treatment - 4 periods of 3 months - 2 group cross-over superiority study.
  All patients will test both insulin treatments (A and F) in alternating periods.
  The patients of group 2 will start with post prandial Faster-acting aspart insulin (FIASP).
  Interventions: Drug: F-A-F-A (FIASP-NovoRapid-FIASP-NovoRapid)

INTERVENTIONS:
Drug: A-F-A-F (NovoRapid-FIASP-NovoRapid-FIASP) — A = pre-prandial aspart insulin (NovoRapid) F = post prandial Faster-acting aspart insulin (FIASP)
  Other Names: All patients will have both treatments: NovoRapid + FIASP
  Arms: Group 1: A-F-A-F
Drug: F-A-F-A (FIASP-NovoRapid-FIASP-NovoRapid) — A = pre-prandial aspart insulin (NovoRapid) F = post prandial Faster-acting aspart insulin (FIASP)
  Other Names: All patients will have both treatments: NovoRapid + FIASP
  Arms: Groupe 2: F-A-F-A

SUMMARY:
Cystic fibrosis related diabetes (CFRD) is a major factor of morbidity and mortality at all disease stages. Insulin deficiency has serious clinical consequences by increasing malnutrition, since protein and lipid catabolism is accelerated in chronic infections. Traditionally, insulin is injected before a meal. Yet, in these patients with highly varied and often staggered nutritional intakes, insulin injection can result in an increased risk of postprandial hypoglycaemia, all the more so as CF patients exhibit decreased glucagon secretion.

Recent progress in the development of new insulins mimicking the physiological secretion more closely has led to ultra-fast insulins (fast aspart), allowing for postprandial hyperglycaemia to be better controlled. In Type 1 diabetics treated with basal-bolus, faster-acting aspart insulin injected after a meal enabled metabolic control comparable to injection of aspart insulin prior to the meal. Fast apart insulin is of particular interest with regard to CFRD, wherein postprandial hyperglycaemia occurs early. In CFRD, these insulins are likewise advantageous in that they can be injected after the meal, thus permitting more flexibility in patients with highly varied diets. Moreover, the insulin dose can be adapted depending on dietary intake, thus preventing hypoglycaemia secondary to highly-varied carbohydrate intakes. Due to its flexibility, this insulin therapy is likely to be better accepted by patients with cystic fibrosis.

DETAILED DESCRIPTION:
The investigators hypothesis that post prandial administration of Insulin faster-acting aspart insulin in patients with CFRD may contribute to a better metabolic control with a decrease of hypoglycaemia and facilitate insulin administration according to the real food intake. The use of Insulin faster-acting aspart insulin will facilitate the functional insulin therapy. More particularly for CF patients, optimization of metabolic control should contribute to maintain a good nutritional status and to slowing the decline of respiratory function and improve the quality of life.

Patients with cystic fibrosis related diabetes and treated by multiple insulin injection (minimal three insulin injection per day or basal bolus insulin regimen) or insulin pump with CGM from over 3 months were included in an open, randomized, two-treatments - 4 periods of 3 months - 2 groups cross-over superiority study. Each group of patients will test both insulin treatments (A = pre prandial Aspart insulin, F = post prandial Faster-acting aspart insulin) in alternating periods with the following sequences: Group 1: A-F-A-F, Group 2: F-A-F-A The patients will be randomized to either one or the other sequence, which defines the groups, and take A or F in each of the 4 periods of the study. Each treatment period will last 3 months.

CGM (free style libre, Abott) will be performed for 2 weeks at baseline and after each 4 months period.

ELIGIBILITY:
Inclusion Criteria:

* Patient with cystic fibrosis related diabetes aged over 10 years (no upper age limite)
* Patient treated by multiple insulin injections (minimal three insulin injections per day or basal bolus insulin regimen) or insulin pump
* Patient with CGM from over 3 months (at the signature of the study's informed consent) or patient not wearing a CGM device, but agreeing a CGM at the inclusion and at the end of each treatment period of 3 months
* Naive patient of Fiasp or patient under Fiasp, having carried out a run-in period of one month with rapid acting insulin treatment
* Affiliated to a social security scheme
* Subject able to understand the objectives and the risks related to the research and to give a dated and signed informed consent
* Subject having been informed of the results of the prior medical examination
* Written informed consent, dated and signed before initiating any trial-related procedure (if the subject is a minor, the consent must be signed by the 2 legal representative and the patient if he/she is able to give consent)

Exclusion Criteria:

* Patient with type 1 or type 2 diabetes
* Patient with cystic fibrosis related diabetes treated with 2 injections / day
* Patient with an HbA1C greater than 12% who demonstrate therapeutic non-compliance
* Patient pregnant (positive urinary pregnancy test) or wishing to pregnancy
* Contraindication to Aspart insulin
* Patient on lung transplant waiting list or transplanted within one year prior to the inclusion visit
* Patient who started treatment with Trikafta® within 3 months prior to the inclusion visit
* Patient who cannot be followed during 12 months
* Subject in exclusion period (determined by previous or current clinical study)
* Impossibility of giving the subject enlightened information (subject in emergency situation, difficulties of understanding, cognitive impairment...)
* Subject under the protection of justice
* Subject under guardianship or curatorship

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2020-08-17 (Actual); Primary Completion 2025-01-20 (Actual); Study Completion 2025-01-20 (Actual)

PRIMARY OUTCOMES:
Change of time in range of blood glucose variation (70-180 mg/dl) versus baseline at the end of each treatment period of 3 months (the last 2 weeks of the period of 3 months) is assessed. | This measurement is assessed at the end of each treatment period of 3 months (the last 2 weeks of the period of 3 months). Month 3, month 6, month 9 and month 12.

SECONDARY OUTCOMES:
Other CGM parameters: mean glucose value per day (mg/dl) | screening(Day 0 to 3 months to Day 0)-Inclusion visit (Day 0)-visit Month 3(3 months after inclusion)-Month 6-Month 9-Month 12
Other CGM parameters: glucose area under the curve for glucose value>180mg/dl - number of glucose values<70 mg/dl-number of glucose values<53mg/dl | screening(Day 0 to 3 months to Day 0)-Inclusion visit (Day 0)-visit Month 3(3 months after inclusion)-Month 6-Month 9-Month 12
Other CGM parameters: time in range of blood glucose >180, >140 <70mg/dl | screening(Day 0 to 3 months to Day 0)-Inclusion visit (Day 0)-visit Month 3(3 months after inclusion)-Month 6-Month 9-Month 12
Hypoglycaemic events experienced by the patient - number of symptomatic hypoglycaemic events under 70 mg/dl par mois - number of major hypoglycaemic events per year - number of nocturnal hypoglycaemic events per month | Inclusion visit (Day0)-visit Month 3(3 months after inclusion visit)-Visit Month 6-Month 9-Month 12
Markers of nutritional status: Body Mass Index (BMI) | visit (Day 0 to 3 months to Day 0-Inclusion visit (Day 0)-visit Month 3 (3 months after inclusion visit)-Visit Month 6-Month 9-Month 12
Markers of nutritional status : bioelectrical impedance - Albumin and Pre albumin | visit (Day 0 to 3 months to Day 0-Inclusion visit (Day 0)-visit Month 3 (3 months after inclusion visit)-Visit Month 6-Month 9-Month 12
Markers of nutritional status : Albumin and Pre albumin (g/l) | visit (Day 0 to 3 months to Day 0-Inclusion visit (Day 0)-visit Month 3 (3 months after inclusion visit)-Visit Month 6-Month 9-Month 12
Markers of metabolic status: HbA1c (mmol/l and %) | screening visit (Day 0 to 3 months to Day 0)-Inclusion visit (Day 0)-visit Month 3 (3 months after inclusion visit)-Visit Month 6-Month 9-Month 12
Markers of metabolic status: daily exogenous need of insulin (UI/day) | screening visit (Day 0 to 3 months to Day 0)-Inclusion visit (Day 0)-visit Month 3 (3 months after inclusion visit)-Visit Month 6-Month 9-Month 12
Assessment of respiratory function parameters : FEV1, CV (L and %) | screening visit (Day 0 to 3 months to Day 0)-Inclusion visit (Day 0)-visit Month 3 (3 months after inclusion visit)-Visit Month 6-Month 9-Month 12
Assessment of respiratory function parameters : O2 saturation (%) | screening visit (Day 0 to 3 months to Day 0)-Inclusion visit (Day 0)-visit Month 3 (3 months after inclusion visit)-Visit Month 6-Month 9-Month 12
Assessment of respiratory function parameters : Number of cures of IV antibiotics per year (collect this information at each visit) | screening visit (Day 0 to 3 months to Day 0)-Inclusion visit (Day 0)-visit Month 3 (3 months after inclusion visit)-Visit Month 6-Month 9-Month 12
Number patients with severe hypoglycaemia and serious adverse events | Inclusion visit (Day 0)-visit Month 3(3 months after inclusion visit)-Visit Month 6-Month 9-Month 12
Other CGM parameters: Time in range of blood glucose 70-140 mg/dl | screening visit (Day 0 to 3 months to Day 0)-Inclusion visit (Day 0)-visit Month 3 (3 months after inclusion visit)-Visit Month 6-Month 9-Month 12

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpitaux Universitaires de Strasbourg, Strasbourg, France

IPD SHARING:
Plan to Share IPD: Undecided